CLINICAL TRIAL: NCT06755853
Title: Scale for the Evaluation of Oral and Pharyngolaryngeal Symptoms After General Anesthesia/A Scale Development Study
Brief Title: Scale for Evaluating Oral and Pharyngolaryngeal Symptoms After General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Fadime Ertural, Principal Investigator, Nuh Naci Yazgan University
Other Study IDs: SEOPSAGA
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: General Anesthesia
Keywords: general anesthesia; Oropharyngeal Symptom; Pharyngolaryngeal Symptom; Scale Development

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients receiving general anesthesia: During general anesthesia, endotracheal intubation or laryngeal mask is usually used to ensure airway patency and prevent aspiration. Both endotracheal tube the researcher will meet face to face with the sample group who volunteered to participate in the study and apply the Informed Consent Form and Sociodemographic Characteristics Form (questions 1-9) before surgery. After surgery, the patient will fill in questions 10-20 of the Sociodemographic Characteristics Form according to the information received from the patient file or healthcare personnel. The Post-General Anesthesia Oral and Pharygolaryngeal Symptoms Assessment Scale will be applied at the 2nd hour after surgery. As a result of the literature review, it was seen that pharyngolaryngeal symptoms were generally evaluated at the 1st, 2nd and 24th hours after surgery.

SUMMARY:
More than 320 million surgical procedures are performed worldwide each year, and most of these procedures are performed under general anesthesia. In such anesthesia practices, patients' airways are usually managed by endotracheal intubation (ETT) or laryngeal mask (LM). These airway management techniques can lead to various pharyngolaryngeal symptoms in the postoperative period. The most common complications include sore throat, hoarseness, difficulty swallowing, and laryngeal injuries. Endotracheal intubation can cause laryngeal injuries, especially during tube placement and removal. These injuries can lead to serious complications such as edema, granuloma, thickening of the vocal cords, subluxation, and nerve palsy. The frequency of postoperative pharyngolaryngeal symptoms varies depending on the type of surgical intervention the patient has undergone, the duration of intubation, and the experience of the operators. Most pharyngolaryngeal injuries are associated with factors such as incorrect placement of the endotracheal tube, overinflation, prolonged indwelling, or incorrect use of the laryngeal mask. However, these symptoms are often considered transient and are often overlooked by patients or healthcare professionals. However, in some cases, long-term functional disorders related to voice, swallowing, and airway patency may develop.

The assessment of pharyngolaryngeal symptoms is critical for more effective management of patients throughout the treatment process and for optimizing their care. Early recognition and management of these symptoms by nurses and other healthcare professionals can reduce complications and increase patient satisfaction.

There is no standard scale in the literature that can assess and classify these symptoms after surgical anesthesia. Existing assessments usually address symptoms separately and are usually performed with subjective measurements. The aim of this study was to develop a scale that can more systematically assess oral and pharyngolaryngeal symptoms such as sore throat, hoarseness, and difficulty swallowing after surgical interventions. Conducting validity and reliability tests of this scale will be an important step in improving patient care during surgical procedures and managing postoperative symptoms more effectively. The aim of this study was to develop a scale to assess pharyngolaryngeal symptoms after general anesthesia and to determine its validity and reliability.

DETAILED DESCRIPTION:
This research is a methodological study conducted to develop a "Post-General Anesthesia Oral and Pharyngolaryngeal Symptoms Assessment Scale".

In order to test the validity and reliability of the Oral and Pharyngolaryngeal Symptoms Evaluation Scale after General Anesthesia, the following application steps will be followed.

Scope Validity The items of the draft scale prepared by the researcher will be asked to be evaluated by experts in the field of Turkish Language and Literature in terms of spelling errors and semantic integrity. Semantic shifts, spelling errors and incorrect expressions will be corrected in line with the feedback given by the experts.

Expert opinion will be sought to ensure the scope validity of the draft scale (each item/question). Scope/content validity is the extent to which the scale as a whole and each item in the scale serves the purpose. Content validity can be evaluated by experts using various techniques. In the Davis technique, items are graded as "appropriate", "item should be slightly revised", "item should be seriously revised" and "item is not appropriate". In this technique, the number of experts who mark the appropriateness of the items and the items should be slightly revised is divided by the total number of experts to obtain the "content validity index" for the item. This value being 0.80 is an acceptable level. A minimum of five and a maximum of 20 experts are sufficient for the Davis technique. Therefore, a minimum of 5 and a maximum of 20 experts will be reached within the scope of the research. For expert opinions, the evaluations of the Anesthesiologist who frequently encounters pharyngolaryngeal symptoms after general anesthesia, surgical nurses in the recovery/recovery unit and academicians in the Surgical Diseases Nursing program will be taken.

Surface Validity A pilot study of the draft scale, whose content validity is provided after the expert opinion, will be conducted. The surface validity of the scale will be ensured with the pilot study. Surface validity is a criterion determined by the researcher himself/herself and the opinions of experts/non-experts on the subject regarding whether a scale measures the structure being investigated. Necessary changes will be made in the meaning and structure in line with the feedback received after the pilot study (Pilot 1 Application). If there is no change in the meaning and structure of the items after the Pilot 1 application, the scale will be applied to a large sample group for the main application of the scale development study. Item analyses will be started with the main application. However, if changes are made to the meaning and structure of the items after the Pilot 1 application, a second expert assessment will be made for content validity.

A pilot study (Pilot 2 application) will be conducted again after the expert opinion is received for the second time. After the integrity of the meaning and structure of the items is determined with the Pilot 2 application, the main application of the scale development study will be conducted. In the main application, the scale will be applied to a large sample group and item analyses will be started and validity-reliability will be tested.

Construct Validity If there is no criterion (reference) to compare the new scale, construct validity should be tested. It provides an explanation of the result obtained from the scale and what this result is related to. It is related to how accurately the prepared scale items measure the specified characteristics. Different researchers point out different methods to evaluate construct validity. The most frequently mentioned of these is factor analysis. Factor Analysis is a construct validity technique used to reveal whether there is a certain order between the responses of the participants to the items in the developed scale. The factor analysis method is used to reveal the basic structure underlying a large number of variables. The aim of this process is to reduce the structure to a smaller number of basic dimensions in order to facilitate the understanding and interpretation of the relationships between a large number of variables thought to be related to each other. Accordingly, Explanatory Factor Analysis (EFA) and Confirmatory Factor Analysis (CFA) will be conducted to ensure the validity of the structure in the research. The acceptable level of factor loading is related to the sample size. For example, if the sample size of a study is at least 350, the acceptable factor loading can be 0.30 or higher. Similarly, for a study with a sample size of at least 200, this value can be 0.40 or higher, and for a study requiring a sample size of at least 120, this value can be 0.50 or higher. If the sample size is 85, the acceptable factor loading should be 0.60 or higher. In a study with a sample size of 60, this value should be 0.70 or higher. Factor loading will be determined according to the sample size and items with low factor loadings will be removed from the draft scale.

Reliability Reliability is the measure of the consistency of the measurement. It is the degree to which the measurement results are free from errors. The measurement results should give similar results when applied in different places. In other words, similar stable results should be obtained in independent measurements. Reliability indicates the extent to which a scale accurately measures the feature it is intended to measure, the productivity and continuity of the scale. For reliability, the test should be repeatable and transferable. Reliability is usually assessed by methods such as internal consistency, parallel (equivalent) forms, test-retest, inter-observer reliability (scoring consistency). Internal consistency and parallel (equivalent) forms methods will be used to test the reliability of the study. When developing a scale, if it consists of questions or items of the same difficulty level and the same content, it can be converted into two equivalent (parallel) forms. In order for the measurements to be equivalent, they must measure the same variable and their means and standard deviations must be equal. In this direction, Visual Analog Scale (VAS) which has a total of 10 symptoms consisting of the same content as the draft scale will be used to determine the parallel form reliability of the draft scale. The correlation between the forms is calculated and interpreted as the reliability coefficient. The internal consistency of a measurement tool is a measure of whether the different items of the tool measure the same concept. There are different calculation and statistical methods for internal consistency analysis. These are: Average of inter-item correlation coefficients, Average of item-total score correlation coefficients, Correlation analysis of binary values and Cronbach's alpha value. The internal consistency of a measurement tool is usually evaluated with statistical methods such as Cronbach's Alpha. With this method, it is determined whether the items are consistent with each other and whether the items measure a hypothetical variable in Likert-type additive scales. High internal consistency coefficients generally above 0.70 indicate that the measurement tool is reliable. The split-half method (split-half method) is also a method used for reliability, in cases where the test can be divided into two halves and a score can be obtained. The method is based on the similarity of the scores obtained from both halves of the sample if the relevant measurement tool is reliable. The method of splitting into two halves can be done as single items-double items or in random order. The correlation between the two halves obtained shows whether it is a reliable measurement tool. The correlation coefficient being above 0.70, that is, being close to 1, shows that the relevant tool is reliable. In the study, Cronbach's Alpha and the relationship coefficient value after the split-half method will be examined to determine reliability. In addition, the average of the Item-total score correlation coefficients will be examined to increase reliability. In this statistical method, it is the correlation of the total scores of the scale with the scores of each item. The average of the item-total score correlation coefficients gives the reliability of the test.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65
* Patients who have received general anesthesia
* Patients who are conscious
* Patients who can communicate verbally
* Patients who volunteer to participate in the study

Exclusion Criteria:

* Patients who received spinal-epidural or regional anesthesia
* Patients who have any discomfort in the oral-pharynx-larynx regions
* Patients who have undergone any surgical intervention in the oral-pharynx-larynx regions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to develop a scale, the sample should be at least 5 times the number of items in the scale and at least 10 times to increase its reliability. For the pilot application, it is sufficient to select 30-50 participants who can represent the target audience. Accordingly, the pilot study will be conducted with 50 people. After the pilot study, construct validity analyses will be conducted using Explanatory Factor Analysis (EFA) and Confirmatory Factor Analysis (CFA) with the remaining items. If there is a sufficiently large sample, it is often recommended to apply EFA to half of the data and CFA to the other half. Therefore, at least five times as many patients as the number of items will be included in the sample group for EFA and at least five times as many patients for CFA.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Draft Scale for Assessing Oral and Pharyngolaryngeal Symptoms After General Anesthesia | Scale Development work takes an average of 2 years
  Since a similar scale to the Post-General Anesthesia Oral and Pharyngolaryngeal Symptom Assessment Scale could not be found, a 46-item oral and pharyngolaryngeal symptom assessment scale created by the researcher based on literature will be used to develop the scale. Reliability and validity studies of the draft scale will be conducted.
Draft Scale for Evaluating Oral and Pharyngolaryngeal Symptoms After General Anesthesia Expert Opinion Evaluation Form | average 2 months
  In order for the draft scale prepared by the researcher to be evaluated by experts, the suitability of the scale items/questions will be measured with the "Expert Opinion Evaluation Form for the Draft Scale for the Evaluation of Oral and Pharyngolaryngeal Symptoms After General Anesthesia".
Vizuel Analog Skalası (VAS) | average 2 years
  The VAS value is determined by measuring the distance between the leftmost end of the scale and the marked point. The scale can be used to evaluate subjective conditions such as pain, anxiety, hunger, thirst, dry mouth, fatigue, weakness, and nausea. The values range from 0 to 10, and higher values indicate an increase in the severity of the symptoms being evaluated. A Visual Analog Scale (VAS) consisting of a total of 10 symptoms (sore throat, dry throat, difficulty swallowing, hoarseness, numbness in the tongue, difficulty speaking, shortness of breath, numbness/abnormal sensation in the throat, change in taste, and dry mouth) consisting of the same content as the prepared draft scale was created. VAS will be used to determine the parallel form reliability of the draft scale.
Sociodemographic Characteristics Form | average 2 years
  The Sociodemographic Characteristics Form created by the researcher consists of a total of 20 questions. The sociodemographic characteristics form was created by the researcher in accordance with the literature. As a result of the literature review, risk factors leading to pharyngolaryngeal injury (gender, age, weight in kilograms, smoking, gastroesophageal reflux history, type and duration of surgical intervention, type of tube used, tube size, difficult intubation, multiple applications of laryngoscope, use of gastric tube, muscle relaxation, use of propofol, postoperative vomiting, pharyngeal aspiration status) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Fadime Ertural, Lecturer, Principal Investigator — Nuh Naci Yazgan University; Salime Mucuk, Prof. Dr., Study Director — TC Erciyes University
Locations (1):
- Erciyes Universty, Kayseri, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I don't want it because the work has not been completed yet.